CLINICAL TRIAL: NCT05212259
Title: A Randomized, Double-Blind, Placebo-controlled, Parallel Design Clinical Study to Evaluate the Effect of Different Doses of UC-II® Supplementation on the Range of Motion & Joint Discomfort in Healthy Subjects
Brief Title: Clinical Study to Evaluate the Effect of Different Doses of UC-II® Supplementation on the Range of Motion & Joint Discomfort in Healthy Subjects
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Vedic Lifesciences Pvt. Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Other
Other Study IDs: LZ/210901/UCII/RMJD
Record Dates: First submitted 2022-01-14; First posted 2022-01-28 (Actual); Last update posted 2022-11-30 (Actual); Status verified 2022-11

CONDITIONS: Joint Pain
MeSH Terms: conditions — Arthralgia | interventions — Collagen Type II; Glucosamine; Chondroitin

STUDY DESIGN:
Intervention Model Description: Randomized, Double-Blind, Placebo-controlled, Parallel Design
Who Masked: Participant, Care Provider, Investigator
Masking Description: Envelope blinding chits
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (5):
- Collagen type II (40 mg/day) (Experimental): 4 capsules per day for 180 days
  Interventions: Drug: Collagen type II (40 mg/day)
- Collagen type II (80 mg/day) (Experimental): 4 capsules per day for 180 days
  Interventions: Drug: Collagen type II (80mg/day)
- Collagen type II (120 mg/day) (Experimental): 4 capsules per day for 180 days
  Interventions: Drug: Collagen type II (120 mg/day)
- Glucosamine Hydrochloride with Chondroitin Sulphate (2700 mg) (Active Comparator): 4 capsules per day for 180 days
  Interventions: Drug: Glucosamine Hydrochloride with Chondroitin Sulphate (2700 mg)
- Placebo (Placebo Comparator): 4 capsules per day for 180 days
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Collagen type II (40 mg/day) — 4 capsules per day
  Arms: Collagen type II (40 mg/day)
Drug: Collagen type II (80mg/day) — 4 capsules per day
  Arms: Collagen type II (80 mg/day)
Drug: Collagen type II (120 mg/day) — 4 capsules per day
  Arms: Collagen type II (120 mg/day)
Drug: Glucosamine Hydrochloride with Chondroitin Sulphate (2700 mg) — 4 capsules per day
  Arms: Glucosamine Hydrochloride with Chondroitin Sulphate (2700 mg)
Drug: Placebo — 4 capsules per day
  Arms: Placebo

SUMMARY:
A Randomized, Double-Blind, Placebo-controlled, Parallel Design Clinical Study to Evaluate the Effect of Different Doses of UC-II® Supplementation on the Range of Motion & Joint Discomfort in Healthy Subjects

ELIGIBILITY:
Inclusion Criteria:

1. Physically active male and female both, aged ≥ 20 to ≤ 65 years with the daily routine of physical exercise (exercise such as walking, jogging, running, cycling, climbing stairs, squatting or any other exercise on investigator's discretion that involves knee joint movement) for at least 3 days a week.
2. Subject with a history of 4-9 months related to knee joint pain aggravation on physical stress.
3. Body mass index (BMI) ≥ 20 and ≤ 29.9 kg/m2.
4. Fasting blood glucose (FBG) ≤ 125 mg/ dl.
5. Subject with self-reported joint pain of ≥ 70 mm on a 100-point VAS scale after 10±2 minutes of walking on a treadmill using modified Naughton protocol.
6. Subject with pain ≤30 mm at rest on Pain VAS
7. Subject not diagnosed as a case of OA / RA confirmed by the American college of rheumatology (ACR) criteria.
8. The subject is willing to complete all the study procedures including study-related questionnaires and tasks, and comply with the study requirements.
9. The subject is willing to abstain from the restricted supplements and medications prior to inclusion and throughout the study period.
10. Subject with the ability to read and provide written, personally signed, and dated informed consent to participate in the study.

Exclusion Criteria:

1. Obese Subject with BMI > 29.9 kg/m2.
2. Subject's inability to complete the exercise protocol of 10±2 minutes at screening.
3. Subject with the clinical diagnosis of any form of joint disease such as Osteoarthritis (OA).
4. Subject with the clinical diagnosis of any form of autoimmune disorder related to the joint such as Rheumatoid arthritis (RA).
5. A subject suffering from Insomnia and restless leg syndrome.
6. Uncontrolled hypertensive defined as subject currently on an anti-hypertensive drug with systolic Blood Pressure ≥ 140 mm Hg and/ or & diastolic blood pressure ≥ 90 mm Hg
7. Uncontrolled diabetics currently on anti-diabetic medication with Fasting blood glucose (FBG) ≥ 126 mg/ dl.
8. Systolic Blood Pressure ≥ 140 mm Hg and/ or & diastolic blood pressure ≥ 90 mm Hg
9. The subject who have been injured near the knee joint region in the past six months.
10. Subject with a history of knee surgery, replacement, or any non-knee surgical procedures that may impact the study outcomes.
11. The subject who have used Intra-articular injections and or steroids for joint health issues in the last six months. The subjects who have undergone a significant cardiovascular event in the past six months.
12. The subject who has undergone a significant cardiovascular event in the past six months.
13. History or presence of clinically significant renal, hepatic, endocrine, biliary, gastrointestinal, pancreatic, or neurological disorders, that in the judgment of the Investigator, would interfere with the subject's ability to provide informed consent, comply with the study protocol (which might confound the interpretation of the study results), or put the subject at undue risk.
14. The subject who have any other chronic disease or condition or inflammatory disease conditions and/ or are using any medication or dietary supplements or ayurvedic medications or topical ointment/oil/gel for joint health that in the judgment of the Investigator would put the subject at unacceptable risk the for the subject in the study or may interfere with evaluations in the study or noncompliance with treatment or visits.
15. Females who are pregnant/planning to be pregnant/lactating or taking any oral contraceptives.
16. The subject who have participated in a study of an investigational product 90 days prior to the screening.
17. Subject with a history of heavy alcohol consumption.
18. Smokers
19. Subject currently on joint health supplements for pain or inflammation.

Ages: 20 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 375 (Estimated)
Dates: Start 2022-10-10 (Actual); Primary Completion 2023-09-15 (Estimated); Study Completion 2023-09-15 (Estimated)

PRIMARY OUTCOMES:
range of motion (active flexion and extension) | from baseline Day 0 to end of study visit day 180
  To evaluate the efficacy of collagen on knee joint flexibility as assessed by the change in the range of motion (active flexion and extension) using goniometry as compared to placebo.

SECONDARY OUTCOMES:
range of motion knee joint flexibility | from baseline (day 0) to end of study visit (day 180)
  Change in the knee joint flexibility (Knee ROM Extension) as assessed by a range of motion (using goniometry) in the Collagen groups versus the other groups
Pain visual analog scale | from baseline (Day 0) to Day 5, 30, 60, 90, 120, 150 and 180
  Knee joint pain as assessed by Pain visual analog scale at the end of the stress exercise in Collagen groups versus the placebo and the Glucosamine & Chondroitin group.
  0 - No pain at all 100 - worst possible pain
Knee injury and Osteoarthritis Outcome Score | from baseline (Day 0) (post-exercise) to follow up visit Day 5, 30, 60, 90, 120, 150 and day 180 (post-exercise)
  Retrospective Joint Discomfort as assessed by the change in the Knee injury and Osteoarthritis Outcome Score as compared in the Collagen groups compared to placebo and Glucosamine & Chondroitin.
  A Likert scale is used and all items have five possible answer options scored from 0 (No problems) to 4 (Extreme problems) and each of the five scores is calculated as the sum of the items included. Scores are transformed to a 0- 100 scale, with zero representing extreme knee problems and 100 representing no knee problems as common in orthopedic scales and generic measures. Scores between 0 and 100 represent the percentage of the total possible score achieved
European Quality of Life Five Dimension five-level | from baseline (Day 0) to the end of the study (day 180)
  Quality of life (QoL) as assessed by change in European Quality of Life Five Dimension five-level score as compared to the change into placebo and Glucosamine & Chondroitin groups Lower level is denoted as 1 and the highest level is denoted as 5

CONTACTS AND LOCATIONS:
Locations (10):
- India (10):
  - HOS Hospital, Ahmedabad, Gujarat
  - Shalby hospital, Surat, Gujarat
  - Aman Hospital and Research Centre, Vadodara, Gujarat
  - BLDEU Hospital and research center, Vijayapura, Karnataka
  - Shree Ashirwad Hospital, Dombivali, Maharashtra
  - Surya Hospital, Nashik, Maharashtra
  - Ranka Hospital, Pune, Maharashtra
  - Jivanrekha Hospital, Pune, Maharashtra
  - BAJ RR Hospital, Thane, Maharashtra
  - Jaipur National University Institute of Medical Sciences and Research Center, Jaipur, Rajasthan

IPD SHARING:
Plan to Share IPD: Undecided